CLINICAL TRIAL: NCT00185133
Title: A Randomized, Double-blind, Placebo-controlled Factorial Study Evaluating the Efficacy and Safety of Co-administration of Olmesartan Medoxomil Plus Amlodipine Compared to Monotherapy in Patients With Mild to Severe Hypertension
Brief Title: Study of Co-administration of Olmesartan Medoxomil Plus Amlodipine in Patients With Mild to Severe Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Reinilde Heyrman, Daiichi Sankyo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS8663-A-U301
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2007-12

CONDITIONS: Hypertension
Keywords: Treatment of high blood pressure in mild to severe hypertensive patients
MeSH Terms: conditions — Hypertension | interventions — Olmesartan Medoxomil; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Olmesartan medoxomil
Drug: Amlodipine

SUMMARY:
This study assesses the efficacy and safety of co-administration of olmesartan medoxomil plus amlodipine in mild to severe hypertensive patients older than 18 years of age

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* 18 years of age or older (20% equal to or older than 65 years)
* With mild to severe hypertension defined as seated diastolic blood pressure of 95-120 mmHg while off any hypertensive medication

Exclusion Criteria:

* Patients should not have serious concomitant conditions that could interfere with the analysis of the results or that could interfere with the well-being of the patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1900
Dates: Start 2005-05; Study Completion 2007-01

PRIMARY OUTCOMES:
Change from baseline in trough seated systolic blood pressure and seated diastolic blood pressure for each treatment arm

SECONDARY OUTCOMES:
To evaluate the number (%) of patients achieving BP goal.
To characterize the pharmacokinetic interactions and the corresponding pharmacodynamic (BP) correlation

CONTACTS AND LOCATIONS:
Locations (139):
- United States (139):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Mobile, Alabama
  - Muscle Shoals, Alabama
  - Tuscumbia, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Anaheim, California
  - Beverly Hills, California
  - Buena Park, California
  - Cypress, California
  - Encino, California
  - Fountain Valley, California
  - La Jolla, California
  - Long Beach, California
  - Los Angeles, California
  - Los Gatos, California
  - Pico Rivera, California
  - Rancho Mirage, California
  - Roseville, California
  - Sacramento, California
  - San Francisco, California
  - Santa Ana, California
  - Spring Valley, California
  - Temecula, California
  - Tustin, California
  - Walnut Creek, California
  - Golden, Colorado
  - Bristol, Connecticut
  - Stratford, Connecticut
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Clearwater, Florida
  - Coral Gables, Florida
  - Daytona Beach, Florida
  - DeLand, Florida
  - Fort Lauderdale, Florida
  - Hialeah, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Kissimmee, Florida
  - Merritt Island, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Palm Harbor, Florida
  - Pembroke Pines, Florida
  - Pinellas Park, Florida
  - Sarasota, Florida
  - Sebastian, Florida
  - Stuart, Florida
  - Tamarac, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Blairsville, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Arkansas City, Kansas
  - Shawnee Mission, Kansas
  - Erlanger, Kentucky
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Auburn, Maine
  - Oxon Hill, Maryland
  - Benzonia, Michigan
  - Cadillac, Michigan
  - Livonia, Michigan
  - Troy, Michigan
  - Brooklyn Center, Minnesota
  - Olive Branch, Mississippi
  - Kansas City, Missouri
  - Butte, Montana
  - Omaha, Nebraska
  - Henderson, Nevada
  - Berlin, New Jersey
  - Elizabeth, New Jersey
  - Hackensack, New Jersey
  - South Bound Brook, New Jersey
  - Turnersville, New Jersey
  - East Syracuse, New York
  - Manlius, New York
  - Rochester, New York
  - Kinston, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Statesville, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Lyndhurst, Ohio
  - Marion, Ohio
  - Mogadore, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Eugene, Oregon
  - Portland, Oregon
  - Beaver, Pennsylvania
  - Bensalem, Pennsylvania
  - Downingtown, Pennsylvania
  - Feasterville, Pennsylvania
  - Fleetwood, Pennsylvania
  - Lansdale, Pennsylvania
  - Philadelphia, Pennsylvania
  - Uniontown, Pennsylvania
  - Cranston, Rhode Island
  - Anderson, South Carolina
  - Charleston, South Carolina
  - Greer, South Carolina
  - Mt. Pleasant, South Carolina
  - Simpsonville, South Carolina
  - Bristol, Tennessee
  - Nashville, Tennessee
  - New Tazewell, Tennessee
  - Arlington, Texas
  - Austin, Texas
  - Carrollton, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Lake Jackson, Texas
  - Midland, Texas
  - New Braunfels, Texas
  - San Angelo, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Burke, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Suffolk, Virginia
  - Lakewood, Washington
  - Olympia, Washington
  - Charleston, West Virginia
  - Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/